CLINICAL TRIAL: NCT05236140
Title: Efficacy of Perineal Electrical Stimulation in Men With Urinary Incontinence After Radical Prostatectomy. A Prospective Randomized Controlled Trial
Brief Title: Electrical Stimulation in Men With Urinary Incontinence After Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hakan Alkan, Clinical Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-151348
Record Dates: First submitted 2022-01-22; First posted 2022-02-11 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Electrical Stimulation
Keywords: perineal electrical stimulation; urinary incontinence; radical prostatectomy
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perineal electrical stimulation (Stimulation group) (Experimental): Perineal electrical stimulation will be performed in lithotomy position via a stimulation device (Enraf Nonius Myomed 632) with perineal surface electrodes. Perineal electrical stimulation will be performed three days a week, 20 minutes a day, a total of 24 sessions for 8 weeks. The stimulation parameters are frequency at 50 Hz, a 5-10s work-rest cycle, and a 300ms pulse width. The symmetric biphasic pulse wave could be delivered over a range of 1-100mA (according to the patient's discomfort level feedback). In this application, three surface electrodes which had 2 cm diameters were used; two electrodes symmetrically at the perianal region (medial to ischial tuberosity); and one electrode at the leg (ground-neutral electrode). Surface electrodes will be used individually for each patient. Perineal electrical stimulation sessions will be performed by an experienced urogynecology rehabilitation nurse.
  Interventions: Device: Perineal electrical stimulation
- Control group (No Intervention): Subjects in the control group will go through baseline assessment and will not receive treatment or instructions to perform pelvic floor exercises at home. After 8 weeks they will be submitted to the final assessment. After the final evaluation, they will be invited to start treatment in the urogynecological rehabilitation unit.

INTERVENTIONS:
Device: Perineal electrical stimulation — Perineal electrical stimulation will be performed in lithotomy position via a stimulation device (Enraf Nonius Myomed 632) with perineal surface electrodes. Perineal electrical stimulation will be performed three days a week, 20 minutes a day, a total of 24 sessions for 8 weeks. The stimulation parameters are frequency at 50 Hz, a 5-10s work-rest cycle, and a 300ms pulse width. The symmetric biphasic pulse wave could be delivered over a range of 1-100mA (according to the patient's discomfort level feedback). In this application, three surface electrodes which had 2 cm diameters were used; two electrodes symmetrically at the perianal region (medial to ischial tuberosity); and one electrode at the leg (ground-neutral electrode). Surface electrodes will be used individually for each patient. Perineal electrical stimulation sessions will be performed by an experienced urogynecology rehabilitation nurse.
  Arms: Perineal electrical stimulation (Stimulation group)

SUMMARY:
Aim: In this study, the investigators aimed to assess the efficacy of perineal electrical stimulation on anxiety, depression, quality of life (QOL), and clinical parameters associated with incontinence in men with urinary incontinence after radical prostatectomy.

Methods: This study is a prospective, randomized controlled trial. The investigators will recruit men who will be referred to the Urogynecological Rehabilitation Unit from other related outpatient clinics with complaints of urinary incontinence after radical prostatectomy. By using a random number generator, men will be randomized into two groups: as follows: perineal electrical stimulation (Group 1), and a control group. A random allocation sequence will be generated at a 1:1 ratio. The primary outcome measure is the continence rates, according to the literature. Furthermore, the severity of incontinence, incontinence episodes, social activity, anxiety, depression as well as QoL were secondary outcome measures. The 24-hour pad test will be carried out to evaluate the severity of incontinence. The Quality of Life-Incontinence Impact Questionnaire (IIQ7) will use to assess specific QoL related to incontinence. The Social Activity Index (SAI) contains, a 10-cm visual analog scale in which men may have problems with participation in social activities (0, impossible to participate;10, no problem to participate) will be used. The Hospital Anxiety and Depression scale (HADS) will use to evaluate the anxiety and depressive symptoms in men with UI after RP in the present study. In addition, treatment satisfaction will be evaluated. Men will evaluate the change in their urinary incontinence on a 5-point Likert scale (5, very satisfied; 1, very unsatisfied)

DETAILED DESCRIPTION:
Group 1: Perineal electrical stimulation (ES) Perineal ES will be performed in lithotomy position via a stimulation device (Enraf Nonius Myomed 632) with perineal surface electrodes. Perineal ES will be performed three days a week, 20 minutes a day, a total of 24 sessions for 8 weeks. The stimulation parameters are frequency at 50 Hz, a 5-10s work-rest cycle and a 300ms pulse width. The symmetric biphasic pulse wave could be delivered over a range of 1-100mA (according to the patient's discomfort level feedback). In this application, three surface electrodes which had 2 cm diameters will be used; two electrodes symmetrically at the perianal region (medial to ischial tuberosity); and one electrode at the leg (ground-neutral electrode). Surface electrodes will be used individually for each patient. Perineal ES sessions will be performed by an experienced urogynecology rehabilitation nurse. Men who missed any therapy sessions for the stimulation group will be excluded from the study.

Group 2: No-treatment (Control group) Subjects in the control group will through baseline assessment and will not receive treatment or instructions to perform pelvic floor exercises at home. After 8 weeks they will submit to the final assessment. After the final evaluation, they will be invited to start treatment in the urogynecological rehabilitation unit.

During the treatment, all men were advised to continue the medical treatment which is not related to incontinence.

Evaluation Parameters The primary outcome measure will be accepted as the continence rates, according to literature. Continence was defined as the loss of 8 grams or less of urine during a 24-hour pad test in patients with urinary incontinence after radical prostatectomy.

Furthermore, the severity of incontinence, incontinence episodes, social activity, anxiety, depression as well as QoL were secondary outcome measures. The 24-hour pad test will be carried out to evaluate the severity of incontinence. It will be used "incontinence episodes" from data collected with a 3-day bladder diary. Patients with a 50% or greater reduction in incontinence episodes will be considered improvement and absence of incontinence was considered dryness. The Quality of Life-Incontinence Impact Questionnaire (IIQ7) will be used to assess specific QoL related to incontinence. The Social Activity Index (SAI) contains, a 10-cm visual analog scale in which men may have problems with participation in social activities (0, impossible to participate;10, no problem to participate) was used. In addition, treatment satisfaction will be evaluated. Men evaluated the change in their UI on a 5-point Likert scale (5, very satisfied; 1, very unsatisfied). The Hospital Anxiety and Depression scale (HADS) will be used to evaluate the anxiety and depressive symptoms in men with UI after RP in the present study. It consists of 14 items and two subscales and has been validated previously. It consists of 14 items each of which is scored 0-3 and two subscales each of which is included seven items and has been validated previously. HADS anxiety (HADS-A) and HADS depression (HADS-D) scores could be derived by summing the subscale items. Higher HADS anxiety and HADS depression scores indicate higher anxiety and depression levels, respectively. Men with HADS anxiety scores ≥8 were classified as having anxiety, while those with HADS depression scores ≥8 were classified as having depression. The Cronbach's alpha coefficient of the HADS was found to be 0.94, indicating good reliability.

All the evaluation tests will be performed by another physician who was blinded to the groups in the initial visit and at the end of the treatment (8th week), except for the continence rate, improvement rate, and the treatment satisfaction parameters which will be evaluated only at the 8th weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. Men with RP with incontinence over >8 gram / 24 hours and no residual cancer after RP on pathological examination.
3. Patients within 2 weeks to 1 year after catheter removal
4. Willingness to complete and do the quality of life scale
5. Understanding procedures, benefits, and possible side effects
6. Being able to give written, informed consent

Exclusion Criteria:

1. UI history before RP
2. History of conservative treatment after RP including ES
3. Prolonged indwelling urethral catheterization (more than 15 days)
4. Previous urological surgery history
5. Transurethral resection of the prostate due to benign prostatic hyperplasia
6. Patients receiving radiotherapy
7. Presence of urethral stricture, and urinary tract infection
8. Heart failure, presence of a pacemaker, implanted defibrillator
9. Use of drugs that may affect bladder function (antimuscarinic, duloxetine, a tricyclic antidepressant, etc.)
10. History of neurogenic bladder, peripheral or central neurological pathology
11. Inability to attend treatment sessions due to distance or physical limitations

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Continence rates | Posttreatment (8th week)
  Continence is defined as the loss of 8 grams or less of urine during a 24-hour pad test in patients with urinary incontinence after radical prostatectomy.

SECONDARY OUTCOMES:
The severity of incontinence | Posttreatment (8th week)
  The 24-hour pad test will be carried out to evaluate the severity of incontinence
Specific quality of life related to incontinence | Posttreatment (8th week)
  The Quality of Life-Incontinence Impact Questionnaire will be used to assess specific QoL related to incontinence (Minumum: 0 maximum:21) higher scores mean worse outcome
The participation in social activities | Posttreatment (8th week)
  The Social Activity Index contains, a 10-cm visual analog scale in which men may have problems with participation in social activities (0, impossible to participate;10, no problem to participate) will be used.
The anxiety and depression | Posttreatment (8th week)
  The Hospital anxiety and depression scale will be used to evaluate the anxiety and depressive symptoms.It consists of 14 items and two subscales and has been validated previously. It consists of 14 items each of which is scored 0-3 and two subscales each of which is included seven items, and has been validated previously. HADS anxiety and HADS depression scores were derived by summing the subscale items. Higher HADS anxiety and HADS depression scores indicate higher anxiety and depression levels, respectively.
treatment satisfaction | Posttreatment (8th week)
  5-point Likert scale higher scores mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Necmettin Yıldız, Prof, Principal Investigator — Pamukkale University
Locations (1):
- Hakan Alkan, Denizli, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu L, Coker AL, Du XL, Cormier JN, Ford CE, Fang S. Long-term survival after radical prostatectomy compared to other treatments in older men with local/regional prostate cancer. J Surg Oncol. 2008 Jun 1;97(7):583-91. doi: 10.1002/jso.21028. PMID 18381603
- [Background] Van Kampen M, De Weerdt W, Van Poppel H, De Ridder D, Feys H, Baert L. Effect of pelvic-floor re-education on duration and degree of incontinence after radical prostatectomy: a randomised controlled trial. Lancet. 2000 Jan 8;355(9198):98-102. doi: 10.1016/S0140-6736(99)03473-X. PMID 10675166
- [Background] Gomes CS, Pedriali FR, Urbano MR, Moreira EH, Averbeck MA, Almeida SHM. The effects of Pilates method on pelvic floor muscle strength in patients with post-prostatectomy urinary incontinence: A randomized clinical trial. Neurourol Urodyn. 2018 Jan;37(1):346-353. doi: 10.1002/nau.23300. Epub 2017 May 2. PMID 28464434
- [Background] Ficarra V, Novara G, Artibani W, Cestari A, Galfano A, Graefen M, Guazzoni G, Guillonneau B, Menon M, Montorsi F, Patel V, Rassweiler J, Van Poppel H. Retropubic, laparoscopic, and robot-assisted radical prostatectomy: a systematic review and cumulative analysis of comparative studies. Eur Urol. 2009 May;55(5):1037-63. doi: 10.1016/j.eururo.2009.01.036. Epub 2009 Jan 25. PMID 19185977
- [Background] Moore KN, Valiquette L, Chetner MP, Byrniak S, Herbison GP. Return to continence after radical retropubic prostatectomy: a randomized trial of verbal and written instructions versus therapist-directed pelvic floor muscle therapy. Urology. 2008 Dec;72(6):1280-6. doi: 10.1016/j.urology.2007.12.034. Epub 2008 Apr 2. PMID 18384853
- [Background] Pedriali FR, Gomes CS, Soares L, Urbano MR, Moreira EC, Averbeck MA, de Almeida SH. Is pilates as effective as conventional pelvic floor muscle exercises in the conservative treatment of post-prostatectomy urinary incontinence? A randomised controlled trial. Neurourol Urodyn. 2016 Jun;35(5):615-21. doi: 10.1002/nau.22761. Epub 2015 Mar 21. PMID 25809925
- [Background] Moore KN, Griffiths D, Hughton A. Urinary incontinence after radical prostatectomy: a randomized controlled trial comparing pelvic muscle exercises with or without electrical stimulation. BJU Int. 1999 Jan;83(1):57-65. doi: 10.1046/j.1464-410x.1999.00894.x. PMID 10233453
- [Background] Hoffmann W, Liedke S, Dombo O, Otto U. [Electrostimulation in therapy of postoperative urinary incontinence. Therapeutic value for quality of life]. Urologe A. 2005 Jan;44(1):33-40. doi: 10.1007/s00120-004-0732-1. German. PMID 15580472
- [Background] Yamanishi T, Mizuno T, Watanabe M, Honda M, Yoshida K. Randomized, placebo controlled study of electrical stimulation with pelvic floor muscle training for severe urinary incontinence after radical prostatectomy. J Urol. 2010 Nov;184(5):2007-12. doi: 10.1016/j.juro.2010.06.103. Epub 2010 Sep 20. PMID 20850831
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Ozlu A, Yildiz N, Oztekin O. Comparison of the efficacy of perineal and intravaginal biofeedback assisted pelvic floor muscle exercises in women with urodynamic stress urinary incontinence. Neurourol Urodyn. 2017 Nov;36(8):2132-2141. doi: 10.1002/nau.23257. Epub 2017 Mar 27. PMID 28345778
- [Background] Moore K, Allen M, Voaklander DC. Pad tests and self-reports of continence in men awaiting radical prostatectomy: establishing baseline norms for males. Neurourol Urodyn. 2004;23(7):623-6. doi: 10.1002/nau.20067. PMID 15382185
- [Background] O'Sullivan R, Karantanis E, Stevermuer TL, Allen W, Moore KH. Definition of mild, moderate and severe incontinence on the 24-hour pad test. BJOG. 2004 Aug;111(8):859-62. doi: 10.1111/j.1471-0528.2004.00211.x. PMID 15270937
- [Derived] Yildiz N, Celen S, Ozlulerden Y, Alkan H. Efficacy of perineal electrical stimulation in men with urinary incontinence after radical prostatectomy. A prospective randomized controlled trial. Neurourol Urodyn. 2023 Jan;42(1):340-348. doi: 10.1002/nau.25096. Epub 2022 Nov 15. PMID 36378836